CLINICAL TRIAL: NCT04724720
Title: A Randomized, Double-Blind, Comparative Trial of the Safety and Efficacy of Famotidine vs Placebo for the Treatment of Non-Hospitalized Symptomatic Adults With COVID-19
Brief Title: Famotidine vs Placebo for the Treatment of Non-Hospitalized Adults With COVID-19
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Cold Spring Harbor Laboratory (Other)
Responsible Party: Principal Investigator, Tobias Janowitz, Study Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-1155
Record Dates: First submitted 2021-01-13; First posted 2021-01-26 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Covid-19
Keywords: Covid-19; Coronavirus; Famotidine; Outpatient; Non-Hospitalized
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Famotidine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind Comparative Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Famotidine (Active Comparator): Participants in this study arm will receive standard of care and prescribed famotidine at 80mg TID for a maximum of 14 days, or until hospital admission.
  Interventions: Drug: Famotidine
- Placebo (Placebo Comparator): Participants in this study arm will receive standard of care and placebo for a maximum of 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famotidine — Standard or care treatment plus prescribed famotidine
  Arms: Famotidine
Drug: Placebo — Standard of care treatment plus placebo
  Arms: Placebo

SUMMARY:
The overall objective of this study is to evaluate the clinical efficacy of oral famotidine in symptomatic non-hospitalized patients with confirmed COVID-19. This study is expected to enroll up to 84 patients with mild to moderate symptoms divided into each of the two study arms. Clinical outcomes of the two treatment arms will be compared. This study will be conducted virtually/remotely.

DETAILED DESCRIPTION:
The outbreak of coronavirus disease 2019 (COVID 19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection was first reported in Wuhan, China, in 31 December 2019 and was declared as a global health emergency on 30 January 2020. Currently, there are no definitive vaccine, therapeutic antibody, or antiviral drug countermeasures currently authorized by the FDA for prevention or treatment of mild to moderate COVID-19 disease.

Famotidine is a histamine-2 receptor antagonist, widely available over-the-counter and at low cost, does not interact with other medications and is safely used for suppression of gastric acid production. This makes it a candidate medication for an ambulatory setting to alleviate the symptoms and shorten the symptomatic period in this population. In a case series of 10 patients with COVID-19 who self-medicated with oral famotidine, significant improvement of symptoms was associated with famotidine use after 24-48 hours. These effects were noted in patients who mostly took doses of 80mg three times daily suggesting that famotidine's action is either through its main known high affinity target, the histamine type 2 receptor or through combined inhibition of histamine receptors. Famotidine may work through reduction of H2R signaling on monocytes with a resulting reduction of cytokine release.

The working hypothesis is that famotidine will be superior to placebo in reducing disease related symptoms in non-hospitalized COVID-19 patients with mild or moderate disease. Patients will be monitored for the duration of the study, as well as be asked to record the severity of their symptoms through a daily questionnaire. Current standard of care (SOC) for patients with mild to moderate COVID-19 in the outpatient setting is to assess risk for severe disease and determine the need for an in-person visit, thromboprophylaxis and adjustment of home medication regimen. If the SOC for COVID-19 patients in the outpatient setting changes during the course of the study, a request will be submitted to modify sections of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
2. Understands and agrees to comply with planned study procedures.
3. Adult ≥18 years of age at time of enrollment.
4. Subject consents to randomization.
5. Subject has confirmed COVID-19 disease < 72 hours prior to randomization.
6. Subject has been experiencing symptoms for >1 day but ≤7 days.
7. Able to use an electronic tablet and Bluetooth devices.
8. Subject has mild to moderate COVID-19 which is defined as (equivalent to 1, 2 on the WHO scale):

   1. Patient does not require immediate admission to the hospital within 24 hrs of initial assessment
   2. Patient does not require supplemental oxygen due to COVID-19
   3. Patient has a score of 2 ("moderate") in at least 3 of the symptoms in the COVID- 19 symptom score

Exclusion Criteria:

1. Any exposure to investigational medications targeting COVID-19 during the present disease. These include recently approves antibodies (passive immunization) for treatment of COVID-19.
2. Use of famotidine within the last 30 days for any indication, e.g. medicating gastric ulcer or recent off label use for COVID-19.
3. Severe COVID-19 disease at time of enrollment requiring admission to hospital.
4. History of Stage 3 severe chronic kidney disease, i.e. eGFR of < 60ml/min.
5. Allergy to famotidine or non-medical ingredients of the study tablet.
6. Known to be immunocompromised by treatment for existing disease due to the immunomodulatory effects of famotidine and therefore possible effects on the pre- existing disease or the immunosuppressive therapy.
7. Patients currently using tizanidine.
8. Documented deficiency of any of the following minerals: Al, Cu, Mn, Fe and Zn.
9. Inability to perform the tasks required for the patient reported outcome measure recordings, including but not restricted to limited language proficiency.
10. Have symptoms of dysphagia or inability to swallow size #000 capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of symptom resolution | Day 28
  Measured by the cumulative incidence of symptom resolution using the "COVID-19 Symptom Score" derived from the answers to a questionnaire based on the NIH endorsed guidelines and the recent FDA guidelines for studying COVID-19 in an outpatient setting. A shorter version has been utilized as a scoring system in the case series of famotidine use in non-hospitalized patients with COVID-19.

SECONDARY OUTCOMES:
Rate of symptom resolution | Day 28
  Assessed by modelling the resolution of cumulative symptoms over time
Cumulative incidence of symptom resolution | Day 60
  Assessed using the "COVID-19 Symptom Score"
Relative change of symptoms | Day 7
  Assessed using the "COVID-19 Symptom Score"
Assessment of Serious Adverse Events | Day 60
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Clinical improvement | Day 28
  Assessed using the 9-point ordinal scale recommended by the WHO for trials enrolling patients with COVID-19.
Improvement in peripheral oxygen saturation | Day 7
  Measured by pulse oximetry in % oxygen saturation.
Mortality | Day 28
  Assessed by counting mortality in each arm
Comparative proportions of hospitalized patients | Day 0-28
  Measured by the proportions of patients having been hospitalized by Day 28.
Change in CRP | Day 7, 14, and 28.
  Measured by CRP [mg/L]
Change in procalcitonin | Day 7, 14, and 28.
  procalcitonin [microg/L]
Change in ferritin | Day 7, 14, and 28.
  ferritin [microg/L]

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Janowitz, MD, PhD, Principal Investigator — Cold Spring Harbor Laboratory
Locations (1):
- Northwell Health, Lake Success, New York, United States

REFERENCES:
- [Background] To KK, Tsang OT, Leung WS, Tam AR, Wu TC, Lung DC, Yip CC, Cai JP, Chan JM, Chik TS, Lau DP, Choi CY, Chen LL, Chan WM, Chan KH, Ip JD, Ng AC, Poon RW, Luo CT, Cheng VC, Chan JF, Hung IF, Chen Z, Chen H, Yuen KY. Temporal profiles of viral load in posterior oropharyngeal saliva samples and serum antibody responses during infection by SARS-CoV-2: an observational cohort study. Lancet Infect Dis. 2020 May;20(5):565-574. doi: 10.1016/S1473-3099(20)30196-1. Epub 2020 Mar 23. PMID 32213337
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Catanzaro M, Fagiani F, Racchi M, Corsini E, Govoni S, Lanni C. Immune response in COVID-19: addressing a pharmacological challenge by targeting pathways triggered by SARS-CoV-2. Signal Transduct Target Ther. 2020 May 29;5(1):84. doi: 10.1038/s41392-020-0191-1. PMID 32467561
- [Background] Wang Y, Zhang D, Du G, Du R, Zhao J, Jin Y, Fu S, Gao L, Cheng Z, Lu Q, Hu Y, Luo G, Wang K, Lu Y, Li H, Wang S, Ruan S, Yang C, Mei C, Wang Y, Ding D, Wu F, Tang X, Ye X, Ye Y, Liu B, Yang J, Yin W, Wang A, Fan G, Zhou F, Liu Z, Gu X, Xu J, Shang L, Zhang Y, Cao L, Guo T, Wan Y, Qin H, Jiang Y, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Remdesivir in adults with severe COVID-19: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2020 May 16;395(10236):1569-1578. doi: 10.1016/S0140-6736(20)31022-9. Epub 2020 Apr 29. PMID 32423584
- [Background] Geleris J, Sun Y, Platt J, Zucker J, Baldwin M, Hripcsak G, Labella A, Manson DK, Kubin C, Barr RG, Sobieszczyk ME, Schluger NW. Observational Study of Hydroxychloroquine in Hospitalized Patients with Covid-19. N Engl J Med. 2020 Jun 18;382(25):2411-2418. doi: 10.1056/NEJMoa2012410. Epub 2020 May 7. PMID 32379955
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Tenforde MW, Kim SS, Lindsell CJ, Billig Rose E, Shapiro NI, Files DC, Gibbs KW, Erickson HL, Steingrub JS, Smithline HA, Gong MN, Aboodi MS, Exline MC, Henning DJ, Wilson JG, Khan A, Qadir N, Brown SM, Peltan ID, Rice TW, Hager DN, Ginde AA, Stubblefield WB, Patel MM, Self WH, Feldstein LR; IVY Network Investigators; CDC COVID-19 Response Team; IVY Network Investigators. Symptom Duration and Risk Factors for Delayed Return to Usual Health Among Outpatients with COVID-19 in a Multistate Health Care Systems Network - United States, March-June 2020. MMWR Morb Mortal Wkly Rep. 2020 Jul 31;69(30):993-998. doi: 10.15585/mmwr.mm6930e1. PMID 32730238
- [Background] Food and Drug Agency Information Sheet on Famotidine, Reference ID: 4280861. 1986. https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/019462s039lbl.pdf.
- [Background] Janowitz T, Gablenz E, Pattinson D, Wang TC, Conigliaro J, Tracey K, Tuveson D. Famotidine use and quantitative symptom tracking for COVID-19 in non-hospitalised patients: a case series. Gut. 2020 Sep;69(9):1592-1597. doi: 10.1136/gutjnl-2020-321852. Epub 2020 Jun 4. PMID 32499303
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Food and Drug Administration. Assessing COVID-19- Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment. (2020).
- [Background] Schulkey CE, Litwin TR, Ellsworth G, Sansbury H, Ahmedani BK, Choi KW, Cronin RM, Kloth Y, Ashbeck AW, Sutherland S, Mapes BM, Begale M, Bhat G, King P, Marginean K, Wolfe KA, Kouame A, Raquel C, Ratsimbazafy F, Bornemeier Z, Neumeier K, Baskir R, Gebo KA, Denny J, Smoller JW, Garriock HA. Design and Implementation of the All of Us Research Program COVID-19 Participant Experience (COPE) Survey. Am J Epidemiol. 2023 Jun 2;192(6):972-986. doi: 10.1093/aje/kwad035. PMID 36799620